CLINICAL TRIAL: NCT01363882
Title: Progression of Respiratory Dysfunction in Amyotrophic Lateral Sclerosis (ALS) Patients: A Comparison of Standard of Practice vs Polysomnography-Directed Nocturnal Non-Invasive Positive Pressure Ventilation
Brief Title: Polysomnography-directed Noninvasive Ventilation in Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment & high rate of failure to complete protocol
Sponsor: Columbia University (Other)
Collaborators: ALS Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAC6753
Record Dates: First submitted 2011-03-28; First posted 2011-06-02 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; Noninvasive Ventilation; Respiratory Dysfunction; Positive Pressure Ventilation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard NIV (Active Comparator): Noninvasive ventilation (NIV) will be initiated and managed as per current standard of practice guided by the American Academy of Neurology (AAN) Practice Parameters (updated in 2009), in all subjects with amyotrophic lateral sclerosis (ALS) and a forced vital capacity of <50% predicted. Sleep studies will be performed at baseline, 2 weeks, 1, 3 and 6 months, but will not influence management of the NIV.
  Interventions: Other: Standard initiation of NIV
- Sleep study titrated NIV (Experimental): ALS subjects in this arm, who are offered NIV for Forced Vital Capacity (FVC) <50% as per AAN Practice Parameters, will have their initial level of NIV determined polysomnographically. They will be followed with sleep studies at 1 month, 3 months and 6 months to reassess NIV efficacy and NIV will be adjusted as necessary to optimize parameters of oxygenation and ventilation.
  Interventions: Other: Sleep study-guided adjustment of NIV

INTERVENTIONS:
Other: Sleep study-guided adjustment of NIV — Sleep studies will be performed at baseline, within 2 weeks to initially titrate NIV, and at 1, 3 and 6 months to assess NIV performance and adjust it as necessary based on oxygenation and ventilation parameters.
  Arms: Sleep study titrated NIV
Other: Standard initiation of NIV — NIV will be initiated and managed as per current standard of practice. Sleep studies will be performed at baseline, 2 weeks, 1, 3 and 6 months to gather data but will not influence NIV management. NIV will be adjusted by a respiratory therapist or the subject's primary physician per waking symptoms.
  Arms: Standard NIV

SUMMARY:
Use of noninvasive ventilation (NIV, also known colloquially as "Bipap") has been associated in some studies with improvement in pulmonary function, quality of life and survival. NIV is typically applied during sleep, and without the benefit of sleep study to determine the optimal settings. The investigators have shown that when NIV is used in this fashion, failure of nocturnal oxygenation and ventilation is prominent. This study is randomizing patients to standard application of NIV vs application guided by use of sleep study data to determine the effect of titrated therapy on pulmonary function, quality of life and survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite Amyotrophic Lateral Sclerosis (ALS) per El Escorial criteria
* Between ages of 18 and 80 yrs old

Exclusion Criteria:

* Inability to clear secretions from the airway
* Life expectancy < 6 months from a comorbid condition
* Dementia sufficient to impair ability to use NIV, perform respiratory muscle pressure testing (PFTs), or complete Health-related Quality of Life (HRQOL) instruments
* Inability to follow up at the ALS Center on a regular basis
* Previously diagnosed obstructive Sleep Apnea

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in spirometric, respiratory muscle strength, and gas exchange measures | Up to 6 months after starting NIV
  FVC (forced vital capacity), FEV1 (forced expiratory volume in 1 second), MIP (maximum inspiratory pressure) and MEP (maximum expiratory pressure

SECONDARY OUTCOMES:
Duration that the Mental Component Summary (MCS) is maintained above 75% of baseline score for the Medical Outcomes Study Health Survey (SF-12) | Up to 6 months after starting NIV
Survival | Up to 6 months after baseline
  Whether sleep study-titrated NIV is associated with trends to improved survival, compared with standardly prescribed (non-titrated) NIV
Nocturnal oxygenation and ventilation | Up to 6 months after starting NIV
  Nadir oxygen saturation, number of oxygen desaturations of 3%/hr (ODI3), % time of sleep spent with oxygen saturation <90%, apnea-hypopnea index, asynchrony index
Modified Borg dyspnea score (see description) | Up to 6 months after baseline
  The Modified Borg Dyspnea Scale is a 10-point Likert scale asking subjects to rate perceived shortness of breath, ranging from 0 (no breathlessness at all) to 10 (maximal breathlessness)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Basner, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States